CLINICAL TRIAL: NCT02355132
Title: Assessing a Medicaid Randomized Insurance Experiment Within Community Clinics
Acronym: AMRIC
Status: Completed | Type: Observational
Sponsor: Oregon Health and Science University (Other)
Collaborators: Kaiser Foundation Hospitals, Center for Health Research (Other); OCHIN, Inc. (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Jennifer E DeVoe, MD DPhil, Associate Professor, Oregon Health and Science University
Other Study IDs: IRB00007327; R01HL107647 (NIH)
Record Dates: First submitted 2015-01-30; First posted 2015-02-04 (Estimated); Last update posted 2016-05-19 (Estimated); Status verified 2015-10

CONDITIONS: Cardiovascular Disease; Cancer
Keywords: Medicaid; public insurance; cardiovascular disease; prevention; community health centers; electronic health records; cancer prevention
MeSH Terms: conditions — Cardiovascular Diseases; Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Insurance Intervention Arm: Oregon OCHIN patients that put their names on the reservation list for the Oregon Experiment and were randomly chosen to apply for insurance coverage via the Oregon Experiment
  Interventions: Other: Insurance Intervention
- Control: Oregon OCHIN patients that put their names on the reservation list for the Oregon Experiment and were not chosen to apply for insurance coverage via the Oregon Experiment

INTERVENTIONS:
Other: Insurance Intervention — Random selection to apply for Medicaid coverage through Oregon Experiment drawings held between March and October 2008
  Groups: Insurance Intervention Arm

SUMMARY:
This study examines the impact of a randomized insurance experiment on preventive services receipt and healthcare utilization in safety net patients using linked public insurance claims and safety net clinics' electronic health record (EHR) data.

DETAILED DESCRIPTION:
In 2008, the Oregon Medicaid program used a "lottery" (Oregon Experiment) to allocate limited insurance resources to low income adults who did not categorically qualify for traditional Medicaid coverage. Thousands were randomly selected to apply for Medicaid; many others were not selected. This "natural policy experiment" is the first population-level randomization of insurance coverage since Rand's 1971-1982 experiment. We will use data from safety net clinics that share a common electronic health record (EHR) operated by OCHIN, a non-profit organization in Portland, Oregon. As one of the nation's largest linked community health center networks, the OCHIN EHR database records nearly all visits to safety net clinics in Oregon with one patient chart linked across >100 community health centers. We will link Medicaid claims data and the OCHIN database to determine patients that had applied to participate in the Oregon Experiment, as well as to determine those that gained insurance via this experiment. We will test the hypothesis that public insurance coverage is associated with higher rates of receiving preventive care services and increased healthcare utilization among persons with a usual source of primary care. To that end, we will analyze preventive care and utilization patterns among the OCHIN clinic patients affected by Oregon's Medicaid Experiment. This study capitalizes on two unique opportunities: an EHR database linking >100 community health centers, and the quasi-experimental design of Oregon's randomized Medicaid experiment.

The specific aims related to the Oregon Experiment are:

1) To compare post-intervention rates of preventive services receipt among OCHIN patients randomized to the Oregon Experiment group (intervention group), compared to those not in the coverage group (comparison group); and 3) To compare post-intervention rates of ambulatory healthcare utilization among OCHIN patients randomized to the Oregon Experiment group (intervention group), compared to those not in the coverage group (comparison group).

ELIGIBILITY:
Inclusion Criteria:

* must have applied for the Oregon Experiment in 2006
* must have been a patient in an Oregon safety net clinic that is part of the OCHIN, Inc network
* for preventive services outcomes only, matched patients had to have been at a clinic with an electronic health record system by 3/11/08

Exclusion Criteria:

* under 19 years of age
* over 64 years of age
* not alive at the end of the 36 month post-period
* unknown/missing gender

Ages: 19 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Adult individuals on the Oregon Experiment 'reservation list' (applied for the Oregon Experiment) linked to individual patients in an Oregon safety net clinic that is part of the OCHIN, Inc network using Link Plus software and demographic variables common to both datasets.
Sampling Method: Non-Probability Sample
Enrollment: 308283 (Actual)
Dates: Start 2011-08; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Preventive service receipt | 36 months post Oregon Experiment selection (post-period)
  Number of patients with receipt of the following preventive services in the post-period (each outcome assessed individually by whether person met age, gender, and diagnosis criteria (if applicable): body mass index, blood pressure, smoking, pap test, mammography, colorectal cancer screening, chlamydia screening, lipid test, flu vaccination, pneumococcal vaccination, HbA1c test, glucose test) using ICD-9-CM diagnosis and procedure codes, CPT and HCPCS codes, LOINC codes, medication codes, relevant code groupings and codes specific to the OCHIN EHR.

SECONDARY OUTCOMES:
Ambulatory healthcare utilization | 36 months post Oregon Experiment selection (post-period)
  Number of visits in the post-period for the following services: total primary care office visits, total behavioral/mental health visits, labs, referrals, immunizations, imaging)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer E DeVoe, MD, DPhil, Principal Investigator — Oregon Health and Science University; Heather Angier, MPH, Study Director — Oregon Health & Science Univerisity

REFERENCES:
- [Derived] Hatch B, Marino M, Killerby M, Angier H, Hoopes M, Bailey SR, Heintzman J, O'Malley JP, DeVoe JE. Medicaid's Impact on Chronic Disease Biomarkers: A Cohort Study of Community Health Center Patients. J Gen Intern Med. 2017 Aug;32(8):940-947. doi: 10.1007/s11606-017-4051-9. Epub 2017 Apr 3. PMID 28374214
- [Derived] Bailey SR, Heintzman JD, Marino M, Hoopes MJ, Hatch BA, Gold R, Cowburn SC, Nelson CA, Angier HE, DeVoe JE. Measuring Preventive Care Delivery: Comparing Rates Across Three Data Sources. Am J Prev Med. 2016 Nov;51(5):752-761. doi: 10.1016/j.amepre.2016.07.004. Epub 2016 Aug 10. PMID 27522472
- [Derived] DeVoe JE, Marino M, Gold R, Hoopes MJ, Cowburn S, O'Malley JP, Heintzman J, Gallia C, McConnell KJ, Nelson CA, Huguet N, Bailey SR. Community Health Center Use After Oregon's Randomized Medicaid Experiment. Ann Fam Med. 2015 Jul-Aug;13(4):312-20. doi: 10.1370/afm.1812. PMID 26195674